CLINICAL TRIAL: NCT02622698
Title: A Randomized Trial of Oral Protein Supplementation Following Non-bariatric Abdominal Surgery
Brief Title: Oral Protein Supplementation Following Non-bariatric Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eisenhower Army Medical Center (U.S. Federal Agency)
Collaborators: Medical Nutrition USA, Inc. (Industry)
Responsible Party: Principal Investigator, Christina Riojas, Christina Riojas, General Surgeon, Eisenhower Army Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 356154
Record Dates: First submitted 2015-12-01; First posted 2015-12-04 (Estimated); Last update posted 2015-12-04 (Estimated); Status verified 2015-12

CONDITIONS: Protein Supplementation

ARMS (2):
- Control (Placebo Comparator): The patients in the control group did not receive any supplementation, and were directed to follow the dietary guidelines of their surgeon.
  Interventions: Other: Placebo
- Treatment (Experimental): Patients were instructed to consume one ounce (containing 16 grams of protein) of the supplement three times daily. No other modifications were made to the patient's diet. Patients were provided with a total of 60 doses, which would last 20 days if they consumed each dose as instructed.
  Interventions: Dietary Supplement: Prostat AWC

INTERVENTIONS:
Dietary Supplement: Prostat AWC — Prostat AWC- patients received protein supplementation after surgery
  Arms: Treatment
Other: Placebo — Placebo- Patients did not take any protein supplementation after surgery
  Other Names: No intervention
  Arms: Control

SUMMARY:
Investigators performed a randomized controlled trial of 62 patients undergoing elective abdominal operations. The treatment group was provided a liquid protein supplement and instructed to take a dose three times daily for the first 20 postoperative days. Investigators followed patients for six months and compared wound healing and changes in weight and laboratory values.

ELIGIBILITY:
Inclusion Criteria:

* patients scheduled to undergo abdominal surgery [cholecystectomy, ventral hernia repair, colectomy, non-bariatric gastric surgery, appendectomy, small bowel resection, lysis of adhesions, liver resection, splenectomy, proctectomy, stoma construction, pancreatic surgery, duodenal surgery, adrenal surgery, renal surgery, or cystectomy]

Exclusion Criteria:

* Age less than 18 years
* Pregnant
* Abdominal surgery within the past 6 months
* Inability to attend follow-up appointments for at least 6 months
* Liver failure (Child-Pugh Class B or C) or kidney failure (glomerular filtration rate (GFR) less than 30).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2011-08; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Change in weight | Preoperative, and then postoperative at 1-2 weeks, 3 weeks, 1 month, 2 months, 3 months, 6 months
  Mean preoperative weight compared to mean postoperative weight at each follow-up appointment. Weight recorded in pounds, subsequent measurements at each postoperative point were normalized to the preoperative weight and reported as a relative percentage of the preoperative weight.

SECONDARY OUTCOMES:
Wound healing | Preoperative, and then postoperative at 1-2 weeks, 3 weeks, 1 month, 2 months, 3 months, 6 months
  Overall wound healing was documented on a scale of 0-2 (0 for unhealed, 1 for partially healed, 2 for completely healed). A wound was considered partially healed if there was any portion of the wound which had epidermal edges that were not in direct contact.
Change in white blood cell count (1x10 3/ uL) | Preoperative, and then postoperative at 1-2 weeks, 3 weeks, 1 month, 2 months, 3 months, 6 months
  Change in white blood cell count relative to preoperative white blood cell count, calculated as absolute change
Change in total protein (g/ dL) | Preoperative, and then postoperative at 1-2 weeks, 3 weeks, 1 month, 2 months, 3 months, 6 months
  Change in total protein at each follow-up point relative to preoperative total protein, calculated as absolute change
Change in albumin (g/ dL) | Preoperative, and then postoperative at 1-2 weeks, 3 weeks, 1 month, 2 months, 3 months, 6 months
  Change in albumin at each follow-up point relative to preoperative albumin, calculated as absolute change
Change in prealbumin (mg/ dL) | Preoperative, and then postoperative at 1-2 weeks, 3 weeks, 1 month, 2 months, 3 months, 6 months
  Change in prealbumin at each follow-up point relative to preoperative prealbumin, calculated as absolute change